CLINICAL TRIAL: NCT05391672
Title: Augmentation of Partial Anterior Cruciate Ligament Tear: Early Results
Acronym: Augmentation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Michael Mikhaeil Attallah Gendy, Michael Mikhaeil, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17101888
Record Dates: First submitted 2022-05-21; First posted 2022-05-26 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: ACL Injury; ACL Augmentation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: prospective case series study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Augmentation group (Other): We will use hamstring graft in which fixation of graft will be by adjustable loop devices for femoral part fixation & Bioscrews +/- staples for tibial part fixation
  Interventions: Procedure: we will do ACL augmentation surgery to the patients who have partial ACL tear

INTERVENTIONS:
Procedure: we will do ACL augmentation surgery to the patients who have partial ACL tear — we will do ACL augmentation surgery to the patients who have ACL partial tear using hamstring graft and fixation of the graft to the femoral part by adjustable loop and tibial part with Bio or peak screws +\- staples.

SUMMARY:
Clinical evaluation for the patients with partial ACL tear who had ACL augmentation

DETAILED DESCRIPTION:
we will do a clinical evaluation depending mainly on IKDC score for patients with partial ACL tear who undergoing ACL augmentation surgery inside Assiut university hospital

ELIGIBILITY:
Inclusion Criteria:

* age from 15 to 50 years old
* Partial ACL tear without any other ligament injury
* with and without meniscal tear
* with and without knee deformity
* recent and chronic injury

Exclusion Criteria:

* younger than 15 and older than 50 y
* multiligament injury
* complete ACL tear
* failed ACL reconstruction or repair

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-09 (Actual); Primary Completion 2026-03-19 (Estimated); Study Completion 2026-03-19 (Estimated)

PRIMARY OUTCOMES:
The main outcome is difference in IKDC scores between the patients | Baseline
  we will evaluate the clinical outcome post operative mainly according to the difference in IKDC score between the patients

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Abd-El Radi, Lecturer, Study Director — Orthopaedic Department , Faculty of medicine, Assiut University
Locations (1):
- Assiyt University, Asyut, Egypt

REFERENCES:
- [Background] Gobbi A, Whyte GP. Long-term Outcomes of Primary Repair of the Anterior Cruciate Ligament Combined With Biologic Healing Augmentation to Treat Incomplete Tears. Am J Sports Med. 2018 Dec;46(14):3368-3377. doi: 10.1177/0363546518805740. Epub 2018 Nov 6. PMID 30398894
- [Background] Dallo I, Chahla J, Mitchell JJ, Pascual-Garrido C, Feagin JA, LaPrade RF. Biologic Approaches for the Treatment of Partial Tears of the Anterior Cruciate Ligament: A Current Concepts Review. Orthop J Sports Med. 2017 Jan 25;5(1):2325967116681724. doi: 10.1177/2325967116681724. eCollection 2017 Jan. PMID 28210653
- [Background] Sabat D, Kumar V. Partial tears of anterior cruciate ligament: Results of single bundle augmentation. Indian J Orthop. 2015 Mar-Apr;49(2):129-35. doi: 10.4103/0019-5413.152394. PMID 26015599
- [Background] Sharp JW, Kani KK, Gee A, Mulcahy H, Chew FS, Porrino J. Anterior cruciate ligament fixation devices: Expected imaging appearance and common complications. Eur J Radiol. 2018 Feb;99:17-27. doi: 10.1016/j.ejrad.2017.12.006. Epub 2017 Dec 9. PMID 29362147